CLINICAL TRIAL: NCT02157896
Title: Dynamic Changes of Vascular Endothelial Growth Factor and Endostatin in Association With Circulating Endothelial Progenitor Cells After Acute Ischemic Stroke
Brief Title: Vascular Endothelial Growth Factor and Endostatin in Angiogenesis After Acute Ischemic Stroke
Status: Completed | Type: Observational
Sponsor: Shanghai 6th People's Hospital (Other)
Responsible Party: Principal Investigator, Hao Chen, Doctor, Shanghai 6th People's Hospital
Other Study IDs: H1583-660110
Record Dates: First submitted 2014-06-04; First posted 2014-06-06 (Estimated); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Acute Ischemic Stroke
Keywords: Acute ischemic stroke; Vascular endothelial growth factor; Endostatin
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Peripheral blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Acute ischemic stroke: Patients who suffered from acute ischemic stroke within 12 hours for the first time before entry into the study, and had a score between 6 and 25 on the National Institutes of Health Stroke Scale (NIHSS).

SUMMARY:
Vascular endothelial growth factor (VEGF) and Endostatin (ES) participate angiogenesis after cerebral ischemia. Circulating endothelial progenitor cells (EPCs) also play a crucial role in neovascularization and tissue repair after acute ischemic stroke (AIS). The investigators sought to compare the expression of VEGF and ES in serum and the circulating EPCs in patients after AIS with that of healthy control subjects. The investigators obtained peripheral blood and serum samples from study subjects. EPCs in blood samples from AIS patients and healthy controls were quantified by flow cytometry 1 day, 3 days, 5 days and 7 days after AIS. VEGF and ES were measured by enzyme linked immunosorbent assay at the same time points. The relation between them and the relation of them to prognosis of such patients with acute ischemic stroke were assessed.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of acute ischemic stroke
* Admission within 12 hours
* National Institutes of Health Stroke Scale score 6-25

Exclusion Criteria:

* Lacunar infarction
* Cerebral hemorrhagic infarction
* Epilepsy or epileptic persons
* History of neurological diseases, myocardial infarction, renal and hepatic abnormalities and metabolic diseases
* Contraindications to antiplatelet treatments
* Died within the first week of hospitalization
* Serial blood samples could not be obtained

Ages: 45 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patient group comprised twenty male and ten female. Their age ranged from 45 to 74 years. Locations of infarct, as evidenced by radiologic and neurologic symptoms or signs, included the territories of the middle cerebral artery (9 cases), the posterior cerebral artery (8 cases) the anterior cerebral artery (6 cases), vertebrobasilar area (5 cases), and watershed area (2 cases with cortical and subcortical low densities crossing typical vascular territories).
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2013-05; Primary Completion 2014-04 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Modified Rankin Scale scores | 3 months
  0 = No symptoms; 1 = No significant disability. Able to carry out all usual activities, despite some symptoms; 2 = Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities; 3 = Moderate
  - Page 3 of 4 [DRAFT] - disability. Requires some help, but able to walk unassisted; 4 = Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted; 5 = Severe disability. Requires constant nursing care and attention, bedridden, incontinent; 6 = Dead.

SECONDARY OUTCOMES:
Glasgow Outcome Scale scores | 3 months
  Glasgow Outcome Scale 1 = death; Glasgow Outcome Scale 2 = vegetative state; Glasgow Outcome Scale 3 = severe neurological deficit; Glasgow Outcome Scale 4 = mild neurological deficit and Glasgow Outcome Scale 5 = premorbid level of functioning or completely recovery.

CONTACTS AND LOCATIONS:
Overall Officials: Lixia Xue, M.D., Ph.D., Study Director — Shanghai 6th People's Hospital
Locations (1):
- Shanghai Sixth People's Hospital, Shanghai, China